# **PrEP-Pro Study Protocol**

## **Official Title**

PrEP-Pro: Adapting a Multicomponent Intervention to Train and Support Providers to Promote PrEP for Adolescent Girls and Young Women in the Deep South

## Institution

University of Alabama at Birmingham

## **Principal Investigators**

Lynn T. Matthews, MD, MPH – University of Alabama at Birmingham Latesha E. Elopre, MD, MSPH – University of Alabama at Birmingham

NCT Number: NCT06487390

Version Date: 3 September 2025

## **Statement of Compliance**

This study will be conducted in compliance with the protocol, Good Clinical Practice (GCP), and all applicable regulatory requirements, including NIH and UAB IRB regulations.

## **Protocol Summary**

This study evaluates PrEP-Pro, a multicomponent training intervention designed to increase PrEP prescribing among Family Medicine (FM) residents providing care to adolescent girls and young women (AGYW) in Alabama. PrEP-Pro integrates provider education, sexual history-taking training, and peer-led support from PrEP Champions. The study will assess feasibility, acceptability, and preliminary effectiveness using a mixed-methods design across up to six FM residency sites.

## **Study Schema**

Phase 1: Development and adaptation with Community and Scientific Advisory Boards' input.

Phase 2a: Pre-test at 2 sites with 2 PrEP Champions and 8–12 residents.

**Phase 2b:** Pilot test at up to 6 sites with 12 Champions and 72 residents over 6 months.

Data collection: Surveys, EMR review, Champion logs, and in-depth interviews.

## **Introduction / Background**

Black adolescent girls and young women (AGYW) in the U.S. South are disproportionately affected by HIV, with rates nearly 9 times higher than White peers. Despite the proven efficacy of pre-exposure prophylaxis (PrEP), uptake among AGYW remains low. Barriers include provider knowledge gaps, lack of sexual history-taking, stigma, and competing clinical demands. Family Medicine (FM) residents are uniquely positioned to deliver preventive care, particularly in underserved areas. PrEP-Pro was developed to address these barriers by training FM residents in HIV prevention and supporting sustainable PrEP prescribing practices.

Additional protocol details are available:

Isehunwa O, Hill S, Menninger A, Hubner B, Krakower D, Long D, Pratt M, Clement M, Wagoner N, Lanzi R, Simpson T, Elopre L, Matthews L. A Multicomponent Intervention to Train and Support Family Medicine Providers to Promote Pre-exposure Prophylaxis (PrEP) for Adolescent Girls and Young Women in the Deep South: Protocol for the PrEP-Pro Study. JMIR Res Protoc 2023;12:e44908. URL: <a href="https://www.researchprotocols.org/2023/1/e44908">https://www.researchprotocols.org/2023/1/e44908</a>. DOI: 10.2196/44908

## **Objectives and Endpoints**

**Primary Objective:** To evaluate the feasibility and acceptability of PrEP-Pro among FM residents.

**Secondary Objectives:** To improve provider knowledge and skills in PrEP prescribing and sexual historytaking; to assess preliminary effectiveness on PrEP prescriptions and HIV/STI testing among AGYW.

**Exploratory Objectives:** To identify multilevel barriers and facilitators of PrEP implementation using COM-B (Capability, Opportunity, Motivation – Behavior) model and CFIR (Consolidated Framework for Implementation Research).

## **Specific Aims**

HIV disproportionately impacts Black adolescent girls and young women (AGYW) in the Deep South. In Alabama, nearly half of PrEP-eligible adolescents are AGYW, yet none in a recent sample of 429 adolescents had been prescribed PrEP. Barriers include limited provider knowledge, infrequent sexual history-taking, and stigma. Family medicine (FM) residents represent a critical workforce to reduce disparities, but current training does not equip them with the skills or motivation to provide PrEP.

**The PrEP-Pro intervention** is a multicomponent training designed to improve PrEP prescribing for AGYW by equipping FM residents with knowledge, skills, and peer support. Guided by the COM-B model and CFIR, PrEP-Pro integrates:

- 1. Education on HIV epidemiology and PrEP.
- 2. Training in sexual history-taking.
- 3. Support from trained peer "PrEP Champions."

## Our Specific Aims are:

**Aim 1:** Adapt PrEP-Pro training materials and tools with input from community and scientific advisory boards, FM residents, and AGYW.

**Aim 2:** Pre-test PrEP-Pro at two FM residency sites to assess feasibility and acceptability, and refine procedures.

**Aim 3:** Conduct a six-month pilot test of PrEP-Pro across up to six FM residency sites to evaluate acceptability, feasibility, and preliminary effectiveness. Identify determinants of implementation at the provider, clinic, and system levels through in-depth interviews and CFIR-guided analysis.

#### Impact:

PrEP-Pro has the potential to transform HIV prevention in the South by training a generation of FM providers to routinely offer PrEP to AGYW, directly addressing a major gap in HIV prevention.

## **Research Strategy**

### Innovation

- Multicomponent intervention: Combines education, skills training, and peer leadership in a single package.
- **Champion model:** Embeds "PrEP Champions" to sustain practice change, a proven implementation strategy adapted here for PrEP.
- **Implementation science framework:** Uses COM-B and CFIR to design, deliver, and evaluate the intervention.

• **Community-engaged design:** CABs of FM residents and AGYW co-develop content, ensuring contextual relevance.

## **Study Design and Procedures**

A mixed-methods, multi-phase implementation science study:

- **Phase 1:** Development and adaptation of PrEP-Pro with CAB/SAB input and FM resident focus groups.
- Phase 2a: Pre-test at two residency training program sites (2 Champions, 8–12 residents).
- Phase 2b: Six-month pilot test at up to six sites (up to 12 Champions, 72 residents).

## **Setting and Sites**

- Cahaba Family Medicine Residency Program
- Montgomery Family Medicine Residency Program
- UAB Huntsville Family Medicine Residency Program
- · Additional sites as identified

Sites serve diverse patient populations with ≥20% Black patients.

## **Participants**

### **Eligibility Criteria:**

- Licensed FM resident (MD or DO).
- Provides care to AGYW in Alabama.
- Practices at clinic with ≥20% Black patient population.
- Willing and able to provide informed consent.

### Sample Size:

- Pre-test: 2 Champions, 8–12 residents.
- Pilot: Up to 12 Champions, ~72 residents.

#### Intervention: PrEP-Pro

## **Core Components:**

- 1. **Provider Education:** HIV epidemiology, PrEP indications/efficacy, prescribing practices.
- 2. **Sexual History Training:** Role-play, scripts, and tools for adolescent-focused sexual history-taking.
- 3. **PrEP Champions:** Peer residents trained more extensively (~4 hours, 3 sessions) to deliver training, provide ongoing support, and sustain intervention at their sites.

#### Materials:

- Training PowerPoints, reference "Badge Buddies," sexual history screening tool, PrEP prescribing guides, and patient-facing handouts.
- Online resource manual (Google Site) with curriculum, troubleshooting guides, and supplemental resources.

## **Study Procedures**

### Phase 2a: Pre-test

1. **Recruitment:** Up to 2 PrEP Champions and 12 residents. Partner program directors nominate potential Champions; those interested contact the study team to complete consent.

Residents invited to participate through training with their residency site. Those interested in participating in the study self-consented and completed the enrollment baseline survey.

### 2. Training PrEP Champions:

- Three sessions (total ~4 hours).
- o Content: HIV epidemiology, PrEP prescribing, sexual history-taking, role-play.
- Delivery training: how to teach peers using standard slides and cases.
- 3. Resident Training: Champions deliver two 1-hour sessions to peers over 1 month.

### 4. Data Collection:

- Pre/post surveys: demographics, PrEP knowledge/attitudes, AIM/IAM/FIM, EPAS.
- o **Champion logs:** time spent, resident contacts, support provided.
- o **IDIs:** up to 9 participants (Champions + residents) provide feedback.
- **EMR review:** de-identified data on PrEP prescriptions, HIV/STI tests (3 months pre- and post-intervention).
- 5. **Refinement:** Content, tools, and procedures adjusted based on pre-test results.

## Phase 2b: Pilot Test

1. **Recruitment:** Up to 12 PrEP Champions and 72 residents. Partner program directors nominate potential Champions; those interested contact the study team to complete consent.

Residents invited to participate through training with their residency site. Those interested in participating in the study self-consented and completed the enrollment baseline survey.

#### 1. Training:

- Champions trained (same as pre-test).
- Champions deliver two 1-hour sessions to peers.
- Fidelity monitored via session observation and audio recording; feedback provided.

## 2. Ongoing Support:

- Champions meet biweekly with site administrators/social workers to troubleshoot insurance and workflow issues.
- Champions log PrEP-related activities and resident contacts.
- Peer Champions connected across sites for shared learning.

#### 3. Data Collection:

- o **Surveys:** at baseline, 3 months, and 6 months.
- Champion logs.
- o **IDIs:** with Champions, residents, AGYW patients, and stakeholders (~50 total).
- EMR review: 6 months pre- and post-intervention, capturing PrEP prescriptions and HIV/STI testing.

#### **Outcomes**

## **Primary Outcomes:**

- Acceptability (AIM, IAM, EPAS).
- Feasibility (FIM, training completion rates, Champion engagement).

## **Secondary Outcomes:**

- Provider PrEP knowledge, attitudes, and willingness to prescribe.
- Frequency of sexual history-taking.
- PrEP prescriptions to AGYW.
- HIV/STI testing for AGYW encounters.

### 3.7 Data Analysis

### Quantitative:

- Descriptive statistics for acceptability/feasibility.
- Pre/post changes in prescribing/testing assessed using Wilcoxon signed-rank,
  McNemar's test, logistic regression, and Poisson regression.
- o Adjustments for provider demographics and site-level factors.

#### Qualitative:

- o Thematic analysis of IDIs guided by COM-B and CFIR.
- Triangulation across surveys, EMR, and interview data.

#### 3.8 Timeline

- Year 1: Intervention adaptation, CAB/SAB input, FGDs.
- Year 2: Pre-test (2 sites), refinement.

• Year 3: Pilot test (up to 6 sites), data collection, analysis.

## **Human Subjects and Oversight**

- **Risk:** Minimal (educational training, surveys, interviews), primarily related to potential discomfort discussing sexual health topics.
- **Benefits:** Participants gain knowledge and skills in HIV prevention; potential improvements in patient care for AGYW.
- **Consent:** Written for residents/Champions; separate consent for interviews.
- **Privacy:** EMR data aggregated and de-identified.
- Compensation: \$50/hour for Champions' additional duties; \$50 for IDI participants.
- **Monitoring:** PI and site investigators review training fidelity, data completeness, and adverse events (none anticipated).

### **Dissemination Plan**

- Findings shared with CAB, SAB, and residency partners.
- Results presented at state, regional, and national conferences.
- Peer-reviewed manuscripts submitted to JMIR, JAIDS, and Journal of Adolescent Health.
- Findings inform NIH proposal for hybrid effectiveness-implementation trial.